CLINICAL TRIAL: NCT04841018
Title: Does Low Dose of Dexamethasone Enhance Analgesic Quality of Caudal Analgesia in Children Undergoing Orchiopexy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2021-0047
Record Dates: First submitted 2021-03-30; First posted 2021-04-12 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Patients With Cryptorchism Who Are Planning to Undergo Orchiopexy
Keywords: caudal block; low dose dexamethasone; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients enrolled are allocated into one of the following two groups: control group (group C) who receive a higher dose of dexamethasone known to enhance the effect of caudal block from previous study (0.5mg/kg) and dexamethasone group (group D) who receive a lower, antiemetic dose of dexamethasone (0.15mg/kg)
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Higher dose of dexamethasone (0.5mg/kg) that is known to enhance the analgesic quality of caudal block from previous study
  Interventions: Drug: High dose dexamethasone
- Dexamethasone (Experimental): Lower, antiemetic dose of dexamethasone (0.15mg/kg)
  Interventions: Drug: Low dose dexamethasone

INTERVENTIONS:
Drug: High dose dexamethasone — After caudal block with 1.2ml/kg of 0.15% ropivacaine, the patient receives 0.5mg/kg of intravenous dexamethasone
  Arms: Control
Drug: Low dose dexamethasone — After caudal block with 1.2ml/kg of 0.15% ropivacaine, the patient receives 0.15mg/kg of intravenous dexamethasone
  Arms: Dexamethasone

SUMMARY:
Caudal block is one of the most effective modalities to reduce pain both during and after the surgery involving areas under the umbilicus. According to previous research, 0.5mg/kg-1.5mg/kg dexamethasone is known to enhance the analgesic quality of caudal block in children. Despite the fact that this high dose of dexamethasone is used to treat airway edema in actual practice and no adverse side effect related to dosage has been reported, it is 3 to 15 times higher than the daily antiemetic dose of dexamethasone that is used in standard care of anesthesia. Therefore, our study aims to assess the effect of the more practical, antiemetic dose of dexamethasone (0.15mg/kg) as an adjuvant to enhance the quality of caudal block through a non-inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

1. Ages from 6 months old to 6 years old
2. Body weight Less than or equal to 16.7kg
3. American Society of Anesthesiologists (ASA) classification I or II
4. Patients receiving orchiopexy under general anesthesia

Exclusion Criteria:

1. Patients with uncorrected cardiac anomalies
2. Patients with vertebral anomalies
3. Diagnosis of diabetes mellitus
4. Diagnosis of adrenal disease
5. Currently on steroid
6. Body temperature above 37.5'C preoperatively
7. Allergy to dexamethasone
8. Laparoscopic surgery

Ages: 6 Months to 6 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 273 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The need for additional analgesics during the first 48 hrs after surgery | Until 48 hours after the surgery
  The child's parent is to be educated prior to the surgery so that when the pain score (FLACC or Wong-Baker Faces Scale) is 4 or above at home, he or she receives an additional acetaminophen. The outcome assessor calls or text messages the parent at 6 hours, 24 hours, and 48 hours after the surgery to assess the need for additional analgesics until 48 hours after the surgery.

SECONDARY OUTCOMES:
Time to the first additional analgesic | Until 48 hours after the surgery
  The outcome assessor calls or text messages the parent at 6 hours, 24 hours, and 48 hours after the surgery to find out when the first acetaminophen was given and how many times in total it was given to the child. Also, the pain scores (FLACC, Wong-Baker Faces Scale, Parent Postoperative Pain Measure) and the satisfaction scores were obtained at each time point.
total number of additional analgesic | Until 48 hours after the surgery
  The outcome assessor calls or text messages the parent at 6 hours, 24 hours, and 48 hours after the surgery to find out when the first acetaminophen was given and how many times in total it was given to the child. Also, the pain scores (FLACC, Wong-Baker Faces Scale, Parent Postoperative Pain Measure) and the satisfaction scores were obtained at each time point.
pain score at each time point | Until 48 hours after the surgery
  The outcome assessor calls or text messages the parent at 6 hours, 24 hours, and 48 hours after the surgery to find out when the first acetaminophen was given and how many times in total it was given to the child. Also, the pain scores (FLACC, Wong-Baker Faces Scale, Parent Postoperative Pain Measure) and the satisfaction scores were obtained at each time point.
scale of satisfaction at each time point | Until 48 hours after the surgery
  The outcome assessor calls or text messages the parent at 6 hours, 24 hours, and 48 hours after the surgery to find out when the first acetaminophen was given and how many times in total it was given to the child. Also, the pain scores (FLACC, Wong-Baker Faces Scale, Parent Postoperative Pain Measure) and the satisfaction scores were obtained at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Rim Lee, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No